CLINICAL TRIAL: NCT06522867
Title: Reliability Evaluation of Intraocular Pressure At Day 1 Following Vitreoretinal Surgery, Comparing Goldmann Applanation Tonometry (Gold Standard) to Icare and Accupen
Brief Title: Evaluation of Intraocular Pressure Following a Vitreoretinal Surgery Using Goldmann Applanation Tonometry, Icare and Accupen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-7144
Record Dates: First submitted 2024-07-16; First posted 2024-07-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-07

CONDITIONS: Intraocular Pressure
Keywords: Intraocular Pressure; Accupen; Icare; Goldmann; vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intraocular pressure measure (Experimental)
  Interventions: Other: Intraocular pressure measure

INTERVENTIONS:
Other: Intraocular pressure measure — The intraocular pressure of the subjects using either the Goldmann applanation tonometer, Icare or Accupen. The order of the measure is randomized.

SUMMARY:
The goal of this prospective controlled study is to measure the reliability of two intraocular pressure (IOP)-measuring instruments in comparison to the gold standard, Goldmann applanation tonometry (GAT) following vitreo-retinal surgery. The main question the current study aims to answer is: are Icare and Accupen as accurate as GAT in measuring IOP one day post eye surgery?

Participants in this study will have their IOP measured by the three different instruments one day post-surgery.

DETAILED DESCRIPTION:
Goldmann applanation tonometry (GAT), used since 1948, is the reference technique for measuring intraocular pressure (IOP) in both healthy patients and those suffering from glaucoma or other eye disorders. However, the use of GAT requires the topical application of fluorescein, local anesthesia, and direct contact with the cornea. In addition to its lack of portability, these characteristics of GAT quickly led clinicians to try to find simpler, less cumbersome, but just as reliable techniques to measure IOP. Among the techniques developed to potentially replace GAT, two portable techniques are particularly easy to use: rebound tonometry (Icare) and portable applanation tonometry (Accupen). Before these techniques are universally and interchangeably used with GAT, their reliability and accuracy must be measured. The majority of studies have evaluated these techniques in glaucomatous or healthy eyes, presenting mixed but promising results. However, only one recent study has evaluated the validity of the two techniques (Icare and TonoPen) in a post-operative context of vitreo-retinal surgery. More data is therefore necessary to come to a definitive conclusion regarding the reliability of Icare and Accupen.

The objective of this study is therefore to determine whether the IOP measured by Accupen and/or Icare is as accurate as that taken by GAT in patients who have undergone vitreo-retinal surgery.

To answer this question, this project will be a prospective controlled study of 67 patients who have undergone vitreo-retinal surgery and who will have their intraocular pressure taken 1 day post-operatively by the 3 instruments mentioned above, in a randomized order. At their 1-day post-operative visit, an ocular medical history will be taken, including the preoperative diagnosis and the type of surgery performed. A resident in ophthalmology at Laval University, will take a series of 2 intraocular pressures with these 3 devices: GAT, Icare, and Accupen and will average for each group.

The project research hypothesis would be that the taking of intraocular pressure by Icare and/or Accupen is as valid as that taken by Goldman's applanation tonometry.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Received a vitreoretinal surgery

Exclusion Criteria:

* Corneal dystrophy
* Corneal surgery (penetrating keratoplasty, DSAEK/DMEK less than 6 months, radial keratotomy)
* Irregular corneal surface
* Active corneal ulcer
* Active epithelial deficit
* Central corneal scarring
* A history of scleral buckle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Absence of difference between intracular pressure measured by devices | at the post-operative visit (1 day after surgery)
  No difference in the intraocular pressure measured by Accupen or Icare compared to Goldmann tonometer.

SECONDARY OUTCOMES:
Reliability and validity of devices at all intracular pressure level | at the post-operative visit (1 day after surgery)
  The devices have the same intraocular pressure measured by Goldmann tonometer at High level of pressure (>24mmHg), moderate level (10-24mmHg) and low level (<10mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Caissie, MD, Principal Investigator — CHU de Québec - Université Laval; Imad E Hachem, MD, Principal Investigator — CHU de Québec - Université Laval
Locations (1):
- Hôpital du Saint-Sacrement, CHU de Québec - Université Laval, Québec, Quebec, Canada